CLINICAL TRIAL: NCT00599924
Title: Phase I Study Of SU011248 In Combination With Oxaliplatin, Leucovorin, And 5-Fluorouracil In Patients With Advanced Solid Malignancies
Brief Title: Study Of Sunitinib Plus FOLFOX In Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181048
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Results first posted 2009-12-09 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Neoplasms; Neoplasms
Keywords: advanced solid tumors,; colorectal cancer,; sunitinib (SUTENT),; FOLFOX
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Sunitinib; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): SU011248 [sunitinib] in combination with FOLFOX; FOLFOX is a chemotherapy regimen that combines oxaliplatin and leucovorin with bolus and infusion 5-FU. The modified FOLFOX 6 (mFOLFOX6) regimen is one of several different regimens of FOLFOX used in clinic, according to different dosages of the 4 drugs. mFOLFOX6 was administered every 2 weeks on Days 1 and 2 of each cycle.
  25, 37.5 and 50 mg/day, oral, administered on an outpatient basis in three different dosing regimens: schedule 2/2 (2 weeks on, 2 weeks off), schedule 4/2 (4 weeks on, 2 weeks off), and continuous daily dosing (every day); FOLFOX will be administered every 2 weeks, using the modified FOLFOX 6 (mFOLFOX6) regimen, consisting of: oxaliplatin 85 mg/m2 + leucovorin 400 mg/m2 as a 2-hr IV infusion; 5-FU 400 mg/m2 IV bolus, followed by - 5-FU 2400 mg/m2 as a 46-hr IV infusion
  Interventions: Drug: sunitinib + FOLFOX

INTERVENTIONS:
Drug: sunitinib + FOLFOX — 37.5 mg sunitinib + modified FOLFOX6 (Schedule 2/2)
  Other Names: Sunitinib malate, SUTENT, mFOLFOX6
Drug: sunitinib + FOLFOX — 50 mg sunitinib + modified FOLFOX6 (Schedule 2/2)
  Other Names: Sunitinib malate, SUTENT, mFOLFOX6
Drug: sunitinib + FOLFOX — 50 mg sunitinib + modified FOLFOX6 ( CRC, only Schedule 2/2)
  Other Names: Sunitinib malate, SUTENT, mFOLFOX6
Drug: sunitinib + FOLFOX — 37.5 mg sunitinib + modified FOLFOX6 (Schedule 4/2)
  Other Names: Sunitinib malate, SUTENT, mFOLFOX6
Drug: sunitinib + FOLFOX — 50 mg sunitinib + modified FOLFOX6 (Schedule 4/2)
  Other Names: Sunitinib malate, SUTENT, mFOLFOX6
Drug: sunitinib + FOLFOX — 37.5 mg sunitinib + modified FOLFOX6 (Continuous Dosing)
  Other Names: Sunitinib malate, SUTENT, mFOLFOX6
Drug: sunitinib + FOLFOX — 25 mg sunitinib + modified FOLFOX6 (Continuous Dosing)
  Other Names: Sunitinib malate, SUTENT, mFOLFOX6

SUMMARY:
This study determined the maximum tolerated dose and safety of SU011248 (sunitinib malate, SUTENT) in combination with FOLFOX [Leucovorin + Fluorouracil (5-FU) + Oxaliplatin]. Three different dosing regimens with starting doses of sunitinib at 37.5 mg/day (Schedule 2/2, Schedule 4/2, and Continuous Dosing) were tested in patients with advanced solid tumors, including colorectal cancer.

DETAILED DESCRIPTION:
Study Design: Treatment, Single Group Assignment (7 cohorts), Open Label, Non-Randomized, Safety Study.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor malignancy (during expansion at the maximum tolerated dose, entry will be limited to patients wtih adenocarcinoma of the colon or rectum)
* Eastern Cooperative Oncology Group (ECOG) 0 or 1

Exclusion Criteria:

* Prior treatment with more than 6 cycles of traditional alkylating agent-based chemotherapy regimens
* Prior treatment with more than 2 cycles of carboplating-based chemotherapy regimens
* For colorectal cancer patients in the expanded cohorts, prior treatment with more than 2 systemic chemotherapy regimens in the metastatic setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181048&StudyName=Study%20Of%20Sunitinib%20Plus%20FOLFOX%20In%20Patients%20With%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Groups:
- 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2); 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2): Schedule 2/2 = Sunitinib administered daily for 2 weeks followed by a 2-week off period. Sunitinib was administered during every other cycle of modified FOLFOX6.
- 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2): CRC = colorectal cancer. Schedule 2/2 = Sunitinib administered daily for 2 weeks followed by a 2-week off period. Sunitinib was administered during every other cycle of modified FOLFOX6.
- 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2); 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2): Schedule 4/2 = Sunitinib administered daily for 4 weeks followed by a 2-week off period, overlapping with 3 cycles of modified FOLFOX6
- 37.5 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing); 25 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing): Continuous Dosing = Sunitinib administered daily for 16 weeks. Off periods and dosage depended on toxicities observed. Sunitinib was administered with modified FOLFOX6.
Period: Overall Study
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing) | 25 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing)
Started | 4 | 9 | 5 | 12 | 9 | 6 | 8
Completed | 1 | 4 | 3 | 4 | 3 | 2 | 3
Not Completed | 3 | 5 | 2 | 8 | 6 | 4 | 5
Not completed — Lack of Efficacy | 3 | 5 | 1 | 2 | 3 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 2 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing) | 25 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing) | Total
Number analyzed (Participants) | 4 | 9 | 5 | 12 | 9 | 6 | 8 | 53
Age, Customized [Number; unit: participants]
  < 65 years | 2 | 6 | 5 | 7 | 6 | 6 | 5 | 37
  > = 65 years | 2 | 3 | 0 | 5 | 3 | 0 | 3 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 2 | 6 | 1 | 2 | 3 | 19
  Male | 3 | 5 | 3 | 6 | 8 | 4 | 5 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: All observed or volunteered AEs and SAEs regardless of treatment group or suspected causal relationship to the investigational product(s) were reported.
Time Frame: up to 20 weeks
Population: Intent to treat (ITT) = all subjects enrolled in the study that received at least one dose of study medication. Subjects who did not complete the follow-up period for dose limiting toxicity assessment because of death from progressive disease or other non-treatment related events were replaced.
Measure: Number; unit: participants
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing) | 25 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing)
Number analyzed (Participants) | 4 | 9 | 5 | 12 | 9 | 6 | 8
participants
  AEs | 4 | 9 | 5 | 12 | 9 | 6 | 8
  SAEs | 0 | 4 | 0 | 7 | 3 | 2 | 4

2. Secondary Outcome: Objective Response (OR)
Description: From the start of treatment until disease progression/recurrence. OR=confirmed Complete Response (CR) or confirmed Partial Response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR = disappearance of all target lesions. CR was confirmed if it persisted on repeat imaging study ≥ 4 weeks after initial documentation of response. PR = ≥ 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. PR was confirmed if it persisted on repeat imaging study ≥ 4 weeks after initial documentation of response.
Time Frame: From start of treatment until Day 8 of Cycles 4 and 8 (2/2 Schedule), Day 8 of Cycles 3 and 6 (4/2 Schedule), and Day 1 of Cycles 3 and 7 (Continuous Dosing)
Population: ITT
Measure: Number; unit: participants
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing) | 25 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing)
Number analyzed (Participants) | 4 | 9 | 5 | 12 | 9 | 6 | 8
participants | 0 | 2 | 0 | 0 | 0 | 0 | 2

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Sunitinib
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: ITT population of subjects who had completed pharmacokinetic (PK) blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2); 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2): Schedule 2/2 = Sunitinib administered daily for 2 weeks followed by a 2-week rest period. Sunitinib was administered during every other cycle of modified FOLFOX6.
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 8
ng/mL
  Cycle 1, Day 14 | 47.13 (13.165) | 61.36 (14.692)
  Cycle 2, Day 1 | 44.95 (14.272) | 60.24 (13.830)

4. Secondary Outcome: Time to Cmax (Tmax) of Sunitinib
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Median (Full Range); unit: hours
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 8
hours
  Cycle 1, Day 14 | 8.00 [6.00 to 10.00] | 10.00 [4.00 to 10.00]
  Cycle 2, Day 1 | 7.00 [6.00 to 24.00] | 8.00 [4.00 to 10.00]

5. Secondary Outcome: Minimum Plasma Concentration (Cmin) of Sunitinib
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 8
ng/mL
  Cycle 1, Day 14 | 34.95 (10.618) | 38.23 (11.629)
  Cycle 2, Day 1 | 30.28 (10.188) | 39.47 (16.632)

6. Secondary Outcome: Clearance (CL/F) of Sunitinib
Description: Drug clearance (CL/F) = dose divided by area under the plasma concentration-time profile from time zero to twenty-four hours.
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 8
L/hr
  Cycle 1, Day 14 | 41.13 (10.104) | 44.29 (5.663)
  Cycle 2, Day 1 | 42.40 (12.700) | 49.44 (16.211)

7. Secondary Outcome: Area Under Plasma Concentration-Time Profile From Time Zero to Twenty-Four Hours Postdose (AUC24) of Sunitinib
Description: AUC24 = Area under the plasma concentration-time profile from time zero (pre-dose) to twenty-four hours. AUC24 was obtained by the Linear/Log trapezoidal method.
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 8
ng*hr/mL
  Cycle 1, Day 14 | 985.43 (251.046) | 1233.73 (322.353)
  Cycle 2, Day 1 | 948.40 (284.871) | 1202.50 (396.337)

8. Secondary Outcome: Terminal Phase Half-Life (t1/2) of Sunitinib
Description: t1/2 = terminal phase half-life. t1/2 was obtained by natural log of 2 (ln2) divided by the rate constant for terminal phase (kel).
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: T1/2 for sunitinib was not calculated due to short observation time.
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Cmax of SU-012662 (Sunitinib's Metabolite)
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 8
ng/mL
  Cycle 1, Day 14 | 18.95 (3.007) | 22.80 (5.189)
  Cycle 2, Day 1 | 18.75 (2.977) | 23.44 (7.094)

10. Secondary Outcome: Tmax of SU-012662 (Sunitinib's Metabolite)
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Median (Full Range); unit: hours
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 8
hours
  Cycle 1, Day 14 | 8.00 [6.00 to 10.00] | 10.00 [0.00 to 24.00]
  Cycle 2, Day 1 | 15.00 [0.00 to 24.00] | 4.00 [2.00 to 24.00]

11. Secondary Outcome: Cmin of SU-012662 (Sunitinib's Metabolite)
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 8
ng/mL
  Cycle 1, Day 14 | 14.45 (3.497) | 15.70 (4.365)
  Cycle 2, Day 1 | 13.59 (4.585) | 17.68 (5.599)

12. Secondary Outcome: AUC24 for SU-012662 (Sunitinib's Metabolite)
Description: as for outcome 7
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose.
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 8
ng*hr/mL
  Cycle 1, Day 14 | 401.51 (63.164) | 468.79 (117.108)
  Cycle 2, Day 1 | 395.82 (66.618) | 495.97 (154.314)

13. Secondary Outcome: CL/F of SU-012662 (Sunitinib's Metabolite)
Description: CL/F = dose divided by area under the plasma concentration-time profile from time zero to twenty-four hours.
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: CL/F was not calculated for SU-012662.
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: T1/2 of SU-012662 (Sunitinib's Metabolite)
Description: t1/2 = terminal phase half-life. t1/2 was obtained by ln2 divided by kel.
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: T1/2 for SU-012662 was not calculated due to short observation time.
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Cmax of Free Platinum
Description: Oxaliplatin was metabolized to platinum and free platinum was measured.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 11
ng/mL
  Cycle 1, Day 1 | 935.25 (442.974) | 634.00 (134.050)
  Cycle 2, Day 1 | 1043.75 (381.656) | 789.43 (239.650)

16. Secondary Outcome: Tmax of Free Platinum
Description: Oxaliplatin was metabolized to platinum and free platinum was measured.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Median (Full Range); unit: hours
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 11
hours
  Cycle 1, Day 1 | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00]
  Cycle 2, Day 1 | 2.00 [2.00 to 2.00] | 2.00 [1.00 to 2.00]

17. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Infinity (AUCinf) for Free Platinum
Description: Oxaliplatin was metabolized to platinum and free platinum was measured. AUCinf = Area under the plasma concentration-time profile from time zero (pre-dose) to infinity. AUCinf was obtained by the Linear/Log trapezoidal method.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 11
ng*hr/mL
  Cycle 1, Day 1 | 7459.28 (2892.442) | 6490.17 (1947.621)
  Cycle 2, Day 1 | 7942.64 (3043.567) | 7092.65 (1906.756)

18. Secondary Outcome: T1/2 for Free Platinum
Description: t1/2 = terminal phase half-life. t1/2 was obtained by ln2 divided by kel. Oxaliplatin was metabolized to platinum and free platinum was measured.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 11
hours
  Cycle 1, Day 1 | 16.15 (3.077) | 15.60 (2.038)
  Cycle 2, Day 1 | 18.55 (5.622) | 31.20 (37.925)

19. Secondary Outcome: Cmax of Total Platinum
Description: Oxaliplatin was metabolized to platinum and total platinum was measured.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 12
ng/mL
  Cycle 1, Day 1 | 2490.00 (748.465) | 2137.14 (415.681)
  Cycle 2, Day 1 | 2905.00 (636.684) | 2641.43 (387.145)

20. Secondary Outcome: Tmax of Total Platinum
Description: Oxaliplatin was metabolized to platinum and total platinum was measured.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Median (Full Range); unit: hours
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 12
hours
  Cycle 1, Day 1 | 2.00 [2.00 to 2.00] | 2.00 [1.00 to 2.00]
  Cycle 2, Day 1 | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 2.00]

21. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Forty-Eight Hours (AUC48) for Total Platinum
Description: Oxaliplatin was metabolized to platinum and total platinum was measured. AUC48 = Area under the plasma concentration-time profile from time zero (pre-dose) to forty-eight hours. AUC48 was obtained by the Linear/Log trapezoidal method.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 12
ng*hr/mL
  Cycle 1, Day 1 | 47264.02 (10509.556) | 43713.95 (5590.750)
  Cycle 2, Day 1 | 56813.62 (11980.029) | 51962.03 (8118.343)

22. Secondary Outcome: Steady State Concentration (Css) of Fluorouracil (5-FU)
Description: Steady state is reached when the amount of drug getting into the system per unit time is equal to the amount of drug cleared from the system.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 12
ng/mL
  Cycle 1, Day 1 | 567.52 (351.207) | 334.26 (89.579)
  Cycle 2, Day 1 | 598.86 (127.635) | 647.32 (284.203)

23. Secondary Outcome: Steady State Clearance (CLss) of 5-FU
Description: CLss was determined by total amount of drug received during infusion or duration of infusion (Ki) divided by Css.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: ITT population of subjects who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 4 | 12
L/hr
  Cycle 1, Day 1 | 284.99 (147.808) | 312.63 (93.563)
  Cycle 2, Day 1 | 174.51 (49.445) | 201.12 (103.534)

24. Secondary Outcome: Area Under the Curve (AUC) of 5-FU
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: AUC for 5-FU was not calculated.
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Cmax of 5-FU
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: Cmax of 5-FU was not calculated.
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: T1/2 of Free Platinum, Total Platinum, and 5-FU
Description: t1/2 = terminal phase half-life. t1/2 was obtained by ln2 divided by kel. Oxaliplatin was metabolized to platinum and free and total platinum were measured.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: T1/2 was not calculated for Free Platinum, Total Platinum, and 5-FU.
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: CL/F of Free Platinum, Total Platinum, and 5-FU
Description: CL/F = dose divided by area under the plasma concentration-time profile from time zero to twenty-four hours.
Time Frame: pre-dose, 1h, 2h, 2 h 5 min, 2h 15 min, 2h 30 min, 2h 45 min, 4h, 6h, 8h, 10h, 24h, and 48h post-dose
Population: CL/F was not calculated for Free Platinum, Total Platinum, and 5-FU.
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Cmin of Free Platinum, Total Platinum, and 5-FU
Time Frame: pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: Cmin was not calculated for Free Platinum, Total Platinum, and 5-FU.
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2)
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Volume Endothelial Transfer Constant (Ktrans) of Tumors in a Selected Group of Subjects Assessed by Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI)
Description: Volume endothelial Ktrans was estimated by fitting the tissue contrast agent time course to the Kety equation (Tofts model for analysis of DCE-MRI data).
Time Frame: Cycle 3 (Day 1), Cycle 3 (Day 8)
Population: No pharmacodynamic assessments were performed due to limited number of DCE-MRI scans collected.
Groups:
- 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2): CRC = colorectal cancer. Schedule 2/2 = Sunitinib administered daily for 2 weeks followed by a 2-week rest period. Sunitinib was administered during every other cycle of modified FOLFOX6.
- 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2); 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2): Schedule 4/2 = Sunitinib administered daily for 4 weeks followed by a 2-week rest period, overlapping with 3 cycles of modified FOLFOX6
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Initial Area Dnder the Contrast Agent Concentration-Time Curve (IAUC) of Tumors in a Selected Group of Subjects Assessed by DCE-MRI
Description: IAUC: The initial area under the curve was estimated by integrating the area under the contrast agent concentration time course for the first 90 seconds after bolus arrival in the tumor.
Time Frame: Cycle 3 (Day 1) and Cycle 3 (Day 8)
Population: No pharmacodynamic assessments were performed due to limited number of DCE-MRI scans collected.
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) | 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) | 37.5 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing) | 25 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing)
Serious Adverse Events (participants affected / at risk) | 0/4 | 4/9 | 0/5 | 7/12 | 3/9 | 2/6 | 4/8
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9 | 5/5 | 12/12 | 9/9 | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) (N=4) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) (N=9) | 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2) (N=5) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) (N=12) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) (N=9) | 37.5 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing) (N=6) | 25 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing) (N=8)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) (N=4) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 2/2) (N=9) | 50 mg Sunitinib + Modified FOLFOX6 (CRC Only, Schedule 2/2) (N=5) | 37.5 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) (N=12) | 50 mg Sunitinib + Modified FOLFOX6 (Schedule 4/2) (N=9) | 37.5 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing) (N=6) | 25 mg Sunitinib + Modified FOLFOX6 (Continuous Dosing) (N=8)
Anaemia (Blood and lymphatic system disorders) | 3 | 7 | 0 | 3 | 3 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 4 | 1 | 0 | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 9 | 3 | 5 | 8 | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 6 | 2 | 2 | 5 | 3 | 3
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 5 | 1 | 2 | 4 | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 5 | 1 | 4 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 4 | 4 | 5 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 2 | 4 | 2 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5 | 4 | 7 | 5 | 4 | 5
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 5 | 4 | 5 | 5 | 5 | 3
Chest pain (General disorders) | 0 | 4 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 1
Fatigue (General disorders) | 2 | 6 | 2 | 6 | 7 | 5 | 4
Mucosal inflammation (General disorders) | 2 | 1 | 3 | 3 | 4 | 2 | 1
Oedema peripheral (General disorders) | 0 | 2 | 0 | 2 | 3 | 2 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 4 | 4 | 0 | 3
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 1 | 2 | 1 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | 1
Aspartate aminotransferase (Investigations) | 0 | 2 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Blood alkaline phosphatase (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 3 | 0 | 0 | 4
Platelet count decreased (Investigations) | 0 | 0 | 1 | 5 | 1 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 4 | 0 | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1 | 4 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 1 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 4 | 2 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 4 | 2 | 1 | 3
Headache (Nervous system disorders) | 0 | 4 | 1 | 2 | 1 | 0 | 2
Hyperaesthesia (Nervous system disorders) | 1 | 1 | 1 | 3 | 1 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1 | 3 | 4 | 1 | 1
Paraesthesia (Nervous system disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 5 | 1 | 1 | 5 | 3 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 3 | 0 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.